CLINICAL TRIAL: NCT05300178
Title: Use of Various Configurations of Different Arterial Grafts in Total Arterial Revascularization
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ahmed samir yussef, teaching assistant, Assiut University
Other Study IDs: coronary revascularization
Record Dates: First submitted 2022-02-24; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Coronary Syndrome; Coronary Disease; Coronary Artery Disease
MeSH Terms: conditions — Angina, Unstable; Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multiple vessel disease: patients with coronary artery disease will be revascularized by using different bypass configuration.
  Interventions: Procedure: coronary artery bypass grafting surgery

INTERVENTIONS:
Procedure: coronary artery bypass grafting surgery — Strategies of Complete Arterial Revascularization THE COMPOSITE TECHNIQUE When the distal RIMA bifurcation cannot loosely reach the LAD, we use the RIMA as a free graft, and a T-shaped , or if more suitable, a Y-shaped anastomosis at the level of the main pulmonary artery, is prepared before connection to cardiopulmonary bypass (CPB) THE CROSS TECHNIQUE The cross arrangement is based on the assumption that patency rates of the right internal mammary artery (RIMA) on the left anterior descending coronary artery (LAD) is similar to that of the left internal mammary artery (LIMA) on the LAD. To improve late survival, every effort should be made to use both IMA grafts for the left system THE IN SITU SEQUENCE When a graft to the posterior wall of the heart is not necessary (the circumflex region), the LIMA is grafted to the left anterior descending and the RIMA to the right coronary artery or its posterior de

SUMMARY:
CABG is a difficult and very critical surgery , it is done to revascularize the myocardium in cases of cardiac ischemia . If the myocardium is still viable in selected patients then it is the treatment of choice with outstanding results . Indications of this operation are more than 50% diameter stenosis of the left main coronary artery, more than 70% diameter stenosis in proximal left anterior descending artery (LAD), more than 70% diameter stenosis in three major coronary vessels, ventricular septal defect related to myocardial infarction , papillary muscle rupture , free wall rupture , ventricular pseudoaneurysm , life-threatening ventricular arrhythmias, and cardiogenic shock. Multiple methods have evolved to achieve the best outcome .The revascularization process depend on two main graft either artery or venous , each has its advantage and disadvantage according to their elasticity , ability to deliver an adequate flow and sustain high blood pressure. Our focus is on the different configuration used for the revascularization by using the artery grafts only due to the superiority of the artery graft in comparison to the venous according to the outcomes and not the feasibility of the technique .It is recommended to begin with internal thoracic artery then saphenous vein if both failed then multiple conduits will be used . Bilateral internal thoracic artery grafting can be an optimal option for coronary artery bypass grafting ,but it's the long-term outcome is still under study.There is no accepted configuration of the anastomosis to be used in the multiple conduits .

ELIGIBILITY:
Inclusion Criteria:

* All patients with multi-coronary vessel disease eligible for CABG surgery .

Exclusion Criteria:

* 1. age more than 70 years 2. diabetic patient 3. single vessel disease 4. associated valvular disease 5. previous open heart surgery 6. hemodynamic unstability 7. Ejection fraction less than (40%)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with multi-coronary vessel disease who are indicated for CABG surgery .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-22 (Estimated); Primary Completion 2022-03-22 (Estimated); Study Completion 2022-03-22 (Estimated)

PRIMARY OUTCOMES:
Effective revascularization. | Changes Baseline perfustion after 3 months by MRI

SECONDARY OUTCOMES:
Number of patient complicated by heart failure | changes in the base line heart rate after 24 hours post-operative

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rocha EAV. Fifty Years of Coronary Artery Bypass Graft Surgery. Braz J Cardiovasc Surg. 2017 Jul-Aug;32(4):II-III. doi: 10.21470/1678-9741-2017-0104. No abstract available. PMID 28977193
- [Background] Garatti A, Castelvecchio S, Canziani A, Santoro T, Menicanti L. CABG in patients with left ventricular dysfunction: indications, techniques and outcomes. Indian J Thorac Cardiovasc Surg. 2018 Dec;34(Suppl 3):279-286. doi: 10.1007/s12055-018-0738-8. Epub 2018 Oct 17. PMID 33060950
- [Background] Amin S, Madsen PL, Werner RS, Krasopoulos G, Taggart DP. Intraoperative flow profiles of arterial and venous bypass grafts to the left coronary territory. Eur J Cardiothorac Surg. 2019 Jul 1;56(1):64-71. doi: 10.1093/ejcts/ezy473. PMID 30715312
- [Background] Kawajiri H, Grau JB, Fortier JH, Glineur D. Bilateral internal thoracic artery grafting: in situ or composite? Ann Cardiothorac Surg. 2018 Sep;7(5):673-680. doi: 10.21037/acs.2018.05.16. PMID 30505752
- [Background] Goldstone AB, Chiu P, Baiocchi M, Wang H, Lingala B, Boyd JH, Woo YJ. Second Arterial Versus Venous Conduits for Multivessel Coronary Artery Bypass Surgery in California. Circulation. 2018 Apr 17;137(16):1698-1707. doi: 10.1161/CIRCULATIONAHA.117.030959. Epub 2017 Dec 14. PMID 29242351